CLINICAL TRIAL: NCT03950557
Title: Post-Operative Cognitive Dysfunction and Delirium After Spinal Surgery: Incidence and Relation With Common Intraoperative Neuromonitoring Data, Blood Pressure Parameters and Concentration of Propofol and Remifentanil Infused With Targeted Controlled Infusion (TCI )
Brief Title: Post Operative Cognitive Dysfunction and Delirium After Spinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Collaborators: Maran Eleonora (Unknown)
Responsible Party: Principal Investigator, Federico Linassi, Principal Investigator, University of Padova
Other Study IDs: FLUO
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Emergence Delirium; Post-Operative Cognitive Dysfunction
Keywords: Infusion pumps; Intraoperative brain monitoring
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this trial is to define if Post-Operative Cognitive Dysfunction and Delirium, detected analyzing changes between pre-operative and post-operative Neurocognitive Test, relate to concentration of effector's site concentration of propofol and remifentanil TCI and to the common intraoperative neuromonitoring values.

DETAILED DESCRIPTION:
Post-Operative Cognitive Dysfunction and Emergence Delirium has not been yet investigated after general anaesthesia with Targeted-Controlled-Infusion (TCI), daily used in the investigator's Hospital to anesthetize patients undergoing spinal surgery. Aim of this trial is to define if neurocognitive tests (Pfeiffer test, Montreal Cognitive Assessment, Trail Making Test A and B, Digit Span Test, Confusion Assessment Method) before and after surgery relate to concentrations at effector's site (Ec) of propofol and remifentanil TCI, the values of Bispectral Index, blood pressure values and usage of drugs to increase arterial blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* General Anaesthesia delivered with Propofol and Remifentanil with Targeted Controlled Infusion
* Surgical duration > 60 minutes

Exclusion Criteria:

* Neurological pathologies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to spinal surgery in general anaesthesia anesthetized with propofol and remifentanil delivered by Targeted-Controlled-Infusion (TCI) pumps. Women will be subjected to neurocognitive tests (MOCA, TMT A and B, DST, Pfeiffer, CAM) the day before surgery, 15 and 60 minutes after awakening (only CAM) and on the first post-operative day. These test will be related to propofol and remifentanil concentrations at effector site during surgery and awakening, to BIS and Entropia values and to intraoperative blood pressure values.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Operative Cognitive Dysfunction in spinal-surgery patients detected with Montreal Cognitive Assessment test | Patients will be subjected to Montreael Cognitive Assessment (MOCA) test one day before surgery and 1 day after surgery. This test has a score ranging from 1 (minimum) to 30 (maximum). Better neurocognitve outcome with higher scores)
  Discover incidence of Post-Operative Cognitive decline analyzing changes in Post-Operative Cognitive Dysfunction changes between Pre-operative Montreal Cognitive Assessment test score and post-operative Montreal Cognitive Assessment test score
Incidence of Post-Operative Cognitive Dysfunction in spinal-surgery patients detected with Trail Making Test A and B | Patients will be subjected to Trail Making Test (TMT) A and B one day before surgery and 1day after surgery. These tests will be evaluated in seconds required to be completed (better neurocognitive outcome with fewer seconds required)
  Discover Post-Operative Cognitive Dysfunction analyzing changes between Pre-operative Trail Making Test A and B test score and post-operative Trail Making Test A and B test score
Incidence of Post-Operative Cognitive Dysfunction in spinal-surgery patients detected with Digit Span Test | Patients will be subjected to DST one day before surgery and 1 day after surgery. Better neurocognitve outcome with higher scores
  Discover Post-Operative Cognitive Dysfunction analyzing changes between Pre-operative Digit Span Test score and post-operative Digit Span Test test score
Incidence of Emergence Delirium in spinal-surgery patients | Patients will be subjected to CAM 15 minutes after the awakening after general anesthesia
  Discover Emergence Delirium analyzing Post-operative Confusion Assessment Method (CAM) delivered 15 minutes after the awakening of patients
Incidence of Emergence Delirium in spinal-surgery patients | Patients will be subjected to CAM 60 minutes after the awakening after general anesthesia
  Discover Emergence Delirium analyzing Post-operative Confusion Assessment Method (CAM) delivered 60 minutes after the awakening of patients

IPD SHARING:
Plan to Share IPD: No